CLINICAL TRIAL: NCT06442605
Title: Clinical Research on the Application of Single-channel Uterine Fibroid Morcellation System in Laparoscopic Myomectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024016
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Leiomyoma, Uterine
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Conventional laparoscopic myomectomy with the use of a single-channel uterine fibroid morcellation system for fragmentation and retrieval of the fibroids.
  Interventions: Device: single-channel uterine fibroid morcellation system
- Control group (Active Comparator): Conventional laparoscopic myomectomy with the use of a multi-channel specimen retrieval bag and a conventional laparoscopic uterine fibroid morcellator for fragmentation and retrieval of the fibroids.
  Interventions: Device: Multi-channel specimen retrieval bag + conventional laparoscopic uterine fibroid morcellator

INTERVENTIONS:
Device: single-channel uterine fibroid morcellation system — Conventional laparoscopic myomectomy is performed with the use of a single-channel uterine fibroid morcellation system for fragmentation and retrieval of the fibroids during the procedure.
  Arms: Experimental group
Device: Multi-channel specimen retrieval bag + conventional laparoscopic uterine fibroid morcellator — In conventional laparoscopic myomectomy, a multi-channel specimen retrieval bag is used during the procedure, along with a conventional laparoscopic uterine fibroid morcellator for fragmentation and retrieval of the fibroids.
  Arms: Control group

SUMMARY:
Research Purpose The purpose of this study is to explore whether the application of a single-channel uterine fibroid morcellation system compared to a multi-channel specimen retrieval bag during laparoscopic myomectomy can shorten the operative time and improve the efficiency of fibroid removal.

Research Design This study is a single-center, randomized, single-blind, 1:1 controlled trial.

Intervention Measures Study participants were randomly assigned in a 1:1 ratio into two groups.

Experimental group: Conventional laparoscopic myomectomy with the use of a single-channel uterine fibroid morcellation system for fragmentation and retrieval of the fibroids.

Control group: Conventional laparoscopic myomectomy with the use of a multi-channel specimen retrieval bag and a conventional laparoscopic uterine fibroid morcellator for fragmentation and retrieval of the fibroids.

Observation Indicators Primary observation indicator: Time required for fibroid fragmentation and retrieval (from the placement of the single-channel uterine fibroid morcellation system or the multi-channel specimen retrieval bag to complete removal from the abdominal cavity).

Secondary observation indicators: Success rate of placement, intraoperative damage and leakage rate, gynecological surgeon satisfaction with the surgery, total weight of retrieved uterine fibroid fragments.

ELIGIBILITY:
Inclusion Criteria:

Patients with uterine fibroids who meet the surgical indications. Patients aged 18 and above but below 45, who strongly request to preserve the uterus.

Patients planning to undergo laparoscopic myomectomy. Those who understand the purpose, procedures, potential risks of this trial, voluntarily participate in this study, and sign the informed consent form.

Exclusion Criteria:

Patients who cannot tolerate laparoscopic surgery due to their overall physical condition.

Patients with multiple fibroids have at least 4 fibroids, with the largest diameter of a single fibroid being equal to or greater than 10cm.

Patients who require surgical procedures other than laparoscopic myomectomy (excluding pelvic adhesion lysis, resection of mesosalpingeal cysts measuring less than 2cm, and superficial intraperitoneal lesions resection/electrocoagulation).

Preoperatively considering the possibility of uterine fibroid malignancy. Patients with preoperative unclear diagnosis, requiring differentiation from ovarian tumors.

Previously undergone lower abdominal or pelvic intraperitoneal surgery, or patients with severe pelvic or abdominal adhesions.

Presence of untreated infectious sexual diseases, including but not limited to vaginitis, cervical inflammatory diseases, and pelvic inflammatory diseases.

Patients who cannot understand the research protocol, cannot cooperate with the research and follow-up, and any other patients that researchers deem unsuitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2025-06-19 (Estimated); Study Completion 2027-06-19 (Estimated)

PRIMARY OUTCOMES:
Time required for fibroid fragmentation and retrieval | intraoperative
  Using a stopwatch, record the time it takes from the placement of the single-channel uterine fibroid morcellation system or the multi-channel specimen retrieval bag until the complete removal of the single-channel uterine fibroid morcellation system or the multi-channel specimen retrieval bag from the abdominal cavity.

CONTACTS AND LOCATIONS:
Overall Officials: Jinyi Tong, Principal Investigator — Affiliated Hangzhou First People's Hospital, School of Medicine, Westlake University
Locations (1):
- Hangzhou First People's Hospita, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
If necessary, other researchers can ask us to share the raw data via email after the results are published.

REFERENCES:
- [Background] Wei Y, Zhou X, Ren QZ, Ma Q, Tao X, Shao M, Jia S. A self-developed contained bag for laparoscopic myomectomy morcellation. Ginekol Pol. 2022;93(8):605-613. doi: 10.5603/GP.a2022.0002. Epub 2022 Mar 22. PMID 35315012
- [Background] Wang W, Liang H, Zhao F, Yu H, Rong C, Feng W, Chen Q, Yang Y, Li Q, Feng D, Dong Y, Xue M, Liang J, Ling B. A Novel Multi-Port Containment System for Laparoscopic Power Morcellation to Prevent Tumoral Spread: A Retrospective Cohort Study. Front Surg. 2022 Feb 3;9:803950. doi: 10.3389/fsurg.2022.803950. eCollection 2022. PMID 35187057
- [Background] Venturella R, Rocca ML, Lico D, La Ferrera N, Cirillo R, Gizzo S, Morelli M, Zupi E, Zullo F. In-bag manual versus uncontained power morcellation for laparoscopic myomectomy: randomized controlled trial. Fertil Steril. 2016 May;105(5):1369-1376. doi: 10.1016/j.fertnstert.2015.12.133. Epub 2016 Jan 19. PMID 26801067